CLINICAL TRIAL: NCT07083271
Title: Evaluation of Financial Toxicity, Caregiver Burden, and Quality of Life in Hospitalized Cancer Patients: A Multicenter Cross-Sectional Observational Study
Brief Title: Financial Toxicity and Quality of Life in Hospitalized Cancer Patients: A Multicenter Study
Acronym: FIN-CARE
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Collaborators: Gazi University (Other); Kocaeli University (Other)
Responsible Party: Principal Investigator, Galip Can Uyar, Principal Investigator, Medical Oncology Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-1249; AEŞH-BADEK-2024-1249 (Other: Etlik City Hospital Scientific Research and Evaluation Committee)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: Financial Toxicity; Cancer Patients
Keywords: Financial Toxicity; Caregiver Burden; Quality of Life; Hospital Anxiety and Depression Scale; EORTC QLQ-C30; Zarit Burden Scale; Supportive Oncology; Psycho-oncology; Cross-sectional study; Cancer-related financial distress
MeSH Terms: conditions — Financial Stress; Caregiver Burden; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized Adult Cancer Patients: Adult cancer patients (≥18 years) who are hospitalized in medical oncology wards and are cognitively capable of completing self-administered questionnaires. Participants will complete validated Turkish versions of the Zarit Caregiver Burden Scale (ZCBS), EORTC QLQ-C30, and Hospital Anxiety and Depression Scale (HADS). Financial toxicity will be evaluated using self-reported data on household income, out-of-pocket treatment expenses, and insurance status. No intervention will be administered.
  Interventions: Other: Administration of validated questionnaires with established Turkish versions

INTERVENTIONS:
Other: Administration of validated questionnaires with established Turkish versions — Participants will complete validated Turkish versions of three self-administered instruments: the Zarit Caregiver Burden Scale (ZCBS), the EORTC QLQ-C30, and the Hospital Anxiety and Depression Scale (HADS). Financial toxicity will be assessed via self-reported socioeconomic data. No clinical, behavioral, or pharmaceutical intervention will be applied.
  Other Names: Psychosocial assessment tools; Self-reported questionnaires

SUMMARY:
This multicenter, cross-sectional observational study aims to evaluate the impact of financial toxicity on caregiver burden, quality of life, and emotional distress among hospitalized adult cancer patients. Participants will complete validated Turkish versions of the Zarit Caregiver Burden Scale, the EORTC QLQ-C30, and the Hospital Anxiety and Depression Scale (HADS). Financial toxicity will be assessed through indicators such as household income, treatment-related costs, and insurance coverage. Informed consent will be obtained from all participants. The study will not impose any financial burden on the participants or the hospital.

Data collection is planned between August 1, 2025 and January 15, 2026 at three tertiary centers: Etlik City Hospital, Gazi University Faculty of Medicine, and Kocaeli University Faculty of Medicine in Turkey. The findings are expected to contribute to the development of targeted support strategies for patients and caregivers in oncology settings.

DETAILED DESCRIPTION:
This is a cross-sectional, multicenter observational study designed to assess the relationship between financial toxicity and caregiver burden, quality of life, and emotional well-being in hospitalized adult patients with cancer. The study population will include patients aged 18 years or older who are hospitalized in oncology wards and mentally capable of completing self-report questionnaires. Exclusion criteria include patients in intensive care units, those with impaired consciousness, severe psychiatric disorders, or those who are pregnant or lactating.

All participants will be asked to complete a battery of validated, Turkish-translated assessment tools covering multiple psychosocial domains:

The Comprehensive Score for Financial Toxicity (COST) will be used to assess perceived financial burden related to cancer care. The Turkish version consists of 11 items, each rated on a 5-point Likert scale. Total scores range from 0 to 44, with lower scores indicating greater financial toxicity. Financial toxicity will be further evaluated using self-reported data on household income, treatment-related out-of-pocket expenses, and insurance coverage.

The Zarit Caregiver Burden Scale (ZCBS) will be administered to evaluate caregiver burden, especially for informal caregivers such as family members. This 22-item instrument is rated on a 5-point Likert scale, generating a total score between 0 and 88. Higher scores reflect greater levels of burden. The Turkish version has demonstrated strong psychometric validity and reliability in oncology and geriatric care settings.

The Hospital Anxiety and Depression Scale (HADS) will be used to evaluate emotional well-being. It comprises 14 items divided into two subscales: anxiety and depression (each 7 items). Each subscale yields a score between 0 and 21; higher scores denote more severe emotional symptoms. The Turkish version has been validated for use in cancer patient populations.

The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) will be applied to assess quality of life across several domains. This 30-item questionnaire includes a global health status scale, five functional scales (physical, role, emotional, cognitive, and social functioning), and nine symptom scales. Each scale is transformed linearly to a 0-100 score, where higher functioning scores indicate better quality of life, and higher symptom scores reflect greater symptom burden. The Turkish version has been culturally and linguistically validated.

All participants will provide written informed consent prior to enrollment. No medical intervention will be applied, and the study will not impose any financial or logistical burden on the patients or the participating institutions. Participation is voluntary, and withdrawal from the study is permitted at any point without consequences. The study protocol has been reviewed and approved by the Scientific Research and Evaluation Board of Etlik City Hospital (BADEK). The study complies with the ethical principles outlined in the Declaration of Helsinki. Data will be anonymized, securely stored, and only used for academic purposes.

Data collection is scheduled to be conducted between August 1, 2025, and January 15, 2026, across three tertiary oncology centers in Turkey: Etlik City Hospital, Gazi University Faculty of Medicine, and Kocaeli University Faculty of Medicine. Data will be analyzed using descriptive statistics, group comparisons (e.g., independent samples t-test, ANOVA), correlation analyses, and multivariable regression modeling to explore the predictors of financial toxicity and associated psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed solid organ malignancy
* Currently receiving inpatient care in the medical oncology service
* Receiving active oncologic treatment and/or supportive care
* Fluent in Turkish (reading and speaking)
* Capable of understanding and answering the administered surveys
* Signed informed consent form

Exclusion Criteria:

* ICU admission at the time of enrollment
* ECOG Performance Status ≥3 or cognitive/clinical condition preventing completion of questionnaires
* Severe cognitive impairment or psychiatric condition interfering with survey participation
* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients with a diagnosis of solid organ malignancy receiving active oncologic treatment or supportive care in the inpatient medical oncology clinic. All participants must be able to provide informed consent and complete validated Turkish questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between Financial Toxicity and Caregiver Burden Among Hospitalized Cancer Patients | At enrollment (single time point assessment during hospitalization)
  This outcome evaluates the correlation between financial toxicity and caregiver burden among hospitalized adult cancer patients. Financial toxicity will be assessed using the validated Turkish version of the Comprehensive Score for Financial Toxicity (COST-FACIT), an 11-item questionnaire rated on a 5-point Likert scale (0 = Not at all, 4 = Very much). Total scores range from 0 to 44; lower scores indicate greater toxicity and financial distress. Caregiver burden will be measured using the validated Turkish version of the Zarit Caregiver Burden Scale (ZCBS), with 22 items rated on a 5-point Likert scale (0 = Never, 4 = Nearly always). Total scores range from 0 to 88; higher scores indicate greater burden and strain. Both scales are widely used in Turkish cancer populations and have shown strong psychometric properties. Correlation between these continuous scale scores will be analyzed using Pearson or Spearman correlation coefficients based on data distribution.

SECONDARY OUTCOMES:
Association Between Financial Toxicity and Emotional Distress | At enrollment (single time point assessment during hospitalization)
  Emotional distress will be assessed using the validated Turkish version of the Hospital Anxiety and Depression Scale (HADS). The outcome will focus on the correlation between financial toxicity parameters (e.g., out-of-pocket expenses, loss of income) and HADS scores. Higher HADS scores indicate increased levels of anxiety and/or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Etlik City Hospital, Department of Medical Oncology
Locations (3):
- Turkey (Türkiye) (3):
  - Kocaeli University, Medical Oncology Department, Kocaeli, İzmit
  - Etlik City Hospital, Medical Oncology Department, Ankara, Yenimahalle
  - Gazi University, Medical Oncology Department, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies and ethical considerations regarding patient confidentiality and data protection. Data use is restricted to the research team listed in the study protocol, and no external data sharing is planned at this stage.